CLINICAL TRIAL: NCT03578497
Title: Effects of Interleukin-1 Receptor Antagonism on Hyperandrogenemia in Women With Polycystic Ovary Syndrome - a Prospective, Interventional, Single-arm, Open-label, Proof-of-concept Study
Brief Title: Effects of Interleukin-1 Receptor Antagonism on Hyperandrogenemia in Women With Polycystic Ovary Syndrome
Acronym: FertIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00780; me16CC6
Record Dates: First submitted 2018-06-21; First posted 2018-07-06 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Interleukin-1 receptor antagonism; Kineret/Anakinra; testosteron; hyperandrogenemia; androstenedione
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IL-1 receptor antagonist Anakinra 100 mg (Experimental): Anakinra (Kineret®; r-metHuIL-1ra, Swedish Orphan Biovitrum AB) is a recombinant, non-glycosylated form of the human IL-1Ra in a 100 mg/ 0.67 ml solution for subcutaneous injection. Anakinra/Kineret® is supplied in single use prefilled glass syringes with 27 gauge needles as a sterile, clear, colorless-to-white, preservative free solution for daily s.c. administration over a time period of 28 days.
  Interventions: Drug: IL-1 receptor antagonist Anakinra

INTERVENTIONS:
Drug: IL-1 receptor antagonist Anakinra — IL-1 receptor antagonist Anakinra is a recombinant, non-glycosylated form of the human IL-1Ra in a 100 mg/ 0.67 ml solution for subcutaneous injection. Standard dosage licensed by the FDA and European Medicines Agency (EMA) is 100 mg Anakinra daily. It is supplied in single use prefilled glass syringes with 27 gauge needles as a sterile, clear, colourless-to-white, preservative free solution for daily s.c. administration.
  Other Names: Kineret

SUMMARY:
A prospective, interventional, open-label, single-arm, proof-of-concept study: 18 women with Polycystic Ovary Syndrome (PCOS) will be treated with 100 mg of Anakinra/Kineret® for 4 weeks. 1 week after last injection patients will have a follow-up and a dexamethasone visit after a dexamethasone suppression test. Goal of this study is to investigate the effect of the Interleukin 1( IL-1) receptor antagonist Anakinra/Kineret® on laboratory and clinical features in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Premenopausal women aged 18 years or older
* Onset of menarche ≥5 years ago
* Diagnosis of PCOS defined by the Rotterdam criteria
* High sensitivity C-reactive protein level ≥1 mg/l
* Follicular phase of menstrual cycle as evident by

  * Serum estradiol level <200 pmol/l AND
  * Serum progesterone level <8 ng/ml
* Willingness to use non-hormonal contraceptive measures adequate to prevent becoming pregnant during the study

Exclusion Criteria:

* Intake of any testosterone level modifying drugs in the 8 weeks prior to study inclusion,
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to Anakinra/Kineret,
* Women who are pregnant or breast feeding,
* Female participants who are ovariectomized or hysterectomised or post-menopausal
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Clinical signs of infection in the week before inclusion or history of a severe infection during the last 2 months,
* Potentially severe immunosuppression or intake of other immunosuppressive drugs
* Severe hematologic disease
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, active carcinoma),
* History of or suspected tuberculosis and/or hepatitis B/C

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Absolute change in fasting serum androstenedione level (nmol/l) from start (baseline, day 1) to one week after treatment start with Anakinra. | 7 days
  Absolute change in fasting serum androstenedione level (nmol/l) from start (baseline, day 1) to one week after treatment start with Anakinra.

SECONDARY OUTCOMES:
Ferriman-Gallwey-score | Day 1 and 28
  Effect of Anakinra/Kineret® on hirsutism by Ferriman-Gallwey-score (representation of hair growth in a male pattern on a woman shown in four different degrees of severity ( 0= no hair growth; 1= light hair growth; 2= moderate hair growth; 4= severe hair growth) in 11 different body parts; namely the upper lip, chin, chest, upper back, lower back, upper abdomen, lower abdomen, arm, forearm, thigh, and lower leg) will be assessed
Sebum production measures | At day 1 and 28
  Effect of Anakinra/Kineret® on sebum production will be assessed with Sebumeter® SM 815, Courage + Khazaka electronic Gesellschaft mit beschränkter Haftung (GmbH)
Self-reported frequency of hair removal (times/week) | At day 1 and 28
  Effect of Anakinra/Kineret® on hirsutism will be assessed
Plewig-Kligman-score | At day 1 and 28
  Effect of Anakinra/Kineret® on acne severity, assessed with Plewig-Kligman score (presentation of comedonal and inflammatory acne severity, separately graded based on the number of lesions and type; lesion counting done at right side of the face, excluding other side, chest and back.
Ovulation and menstruation rates [%] | Between day 1 and day 35
  Effect of Anakinra/Kineret® on ovulation and menstruation rates will be assessed
Estradiol (pmol/l), free testosterone (nmol/l), total testosterone (nmol/l), sex hormone-binding globulin (SHBG) [nmol/l], Anti-Muellerian Hormone [pmol/l], dehydroepiandrosterone (DHEA) [nmol/l]), basal cortisol (nmol/l) | Day 1, 7, 14, 21, 28 and 35
  Effect of Anakinra/Kineret® on peripheral (sexual) hormones will be assessed
Fasting glucose (mmol/l), homeostatic model of assessment of insulin resistance (HOMA-IR) | At day 1, 7, 14, 21, 28 and 35
  Effect of Anakinra/Kineret® on glucose metabolism will be assessed
Pituitary hormones (luteinizing hormone (LH), follicle stimulating hormone (FSH), adrenocorticotropic hormone (ACTH) [IU/L]) | Day 1, 7, 14, 21, 28 and 35
  Effect of Anakinra/Kineret® on the pituitary-gonadal axis will be assessed
Treatment response according to a Dexamethasone suppression test | At days 35 and 36
  Dexamethasone suppression test will be evaluated as a predictor for treatment response
inflammatory marker white blood cell count [x109/l], | Day 1, 7, 14, 21, 28 and 35
  Time course of inflammatory marker white blood cell count [x109/l] will be assessed
inflammatory marker C reactive protein (CRP) [mg/l] | Day 1, 7, 14, 21, 28 and 35
  Time course of inflammatory marker CRP [mg/l] will be assessed
inflammatory marker IL-6 [pg/ml] | Day 1 and 28
  Time course of inflammatory marker IL-6 [pg/ml] will be assessed
inflammatory marker IL-1Ra [pg/ml] | Day 1, 7, 14, 21, 28 and 35
  Time course of inflammatory marker IL-1Ra [pg/ml] will be assessed
Change in androstenedione level (nmol/l) from start (baseline, day 1) to days 14, 21, 28, and 35 after treatment start with Anakinra. | Days 14, 21, 28, and 35 after treatment start with Anakinra
  Change in androstenedione level (nmol/l) from start (baseline, day 1) to days 14, 21, 28, and 35 after treatment start with Anakinra.
Change in 11-oxygenated androgens (e.g. 11-ketotestosterone, 11-ketoandrostenedione, 11β-hydroxytestosterone, 11β-hydroxyandrostenedione [nmol/l]) on days 7, 14, 28, and 35 after treatment start with Anakinra | Days 7, 14, 28, and 35 after treatment start with Anakinra
  Change in 11-oxygenated androgens (e.g. 11-ketotestosterone, 11-ketoandrostenedione, 11β-hydroxytestosterone, 11β-hydroxyandrostenedione [nmol/l]) on days 7, 14, 28, and 35 after treatment start with Anakinra

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Dep. of Endocrinology, Diabetes and Metabolism
Locations (1):
- University Hospital Basel Endocrinology, Diabetes and Metabolism, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No